CLINICAL TRIAL: NCT00005588
Title: Standardization of Breast Radiotherapy: Trial A - A Randomized Comparison of Fractionation Regimens After Local Excision or Mastectomy in Women With Early Stage Breast Cancer
Brief Title: Radiation Therapy After Surgery in Treating Women With Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067662; STMG-STARTA; EU-99014
Record Dates: First submitted 2000-05-02; First posted 2003-05-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of radiation therapy is more effective following surgery for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of radiation therapy following surgery in treating women who have early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the benefits of radiotherapy schedules using fraction sizes larger than 2.0 Gy in terms of normal tissue responses, local-regional tumor control, quality of life, and economic consequences in women prescribed postoperative radiotherapy for early stage breast cancer.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, type of surgery (mastectomy vs local excision), and breast boost (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive radiotherapy 5 times a week for 5 weeks for a total dose of 50 Gy.
* Arm II: Patients receive radiotherapy 5 times a fortnight (i.e., Monday/Wednesday/Friday/Tuesday/Thursday/Monday, etc.) for 13 fractions over 5 weeks for a total dose of 41.6 Gy.
* Arm III: Patients receive radiotherapy as in arm II for a total dose of 39 Gy. A breast boost is recommended in all arms for patients with microscopic evidence of invasive or in situ cancer at, or within 1 mm of, a resection margin. These patients receive radiotherapy for 5 fractions in 1 week for a total boost dose of 10 Gy.

Quality of life is assessed at baseline and then at 6, 12, 24, and 60 months.

Patients are followed annually for up to 20 years.

PROJECTED ACCRUAL: A total of 2,010 patients (670 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive unilateral breast cancer that is considered operable

  * T1-3, N0-1, M0 at presentation
* Complete macroscopic excision of tumor by breast conserving surgery or mastectomy
* No immediate breast reconstruction
* No requirement for axillary radiotherapy after greater than a Level 1 axillary dissection or after greater than 10 lymph nodes have been removed
* Not enrolled on SECRAB or OSCAR trials
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

* Prior neoadjuvant, or primary medical, therapy allowed provided subsequent surgery confirms complete macroscopic excision of residual primary tumor

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 weeks since prior cytotoxic agents
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (32):
- United Kingdom (32):
  - Royal Sussex County Hospital, Brighton, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Cheltenham General Hospital, Cheltenham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Royal Surrey County Hospital, Guildford, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - University Hospitals of Leicester, Leicester, England
  - Guy's and St. Thomas' Hospitals Trust, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - South Tees Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - King Edward VII Hospital, Midhurst, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Royal Berkshire Hospital, Reading, England
  - Oldchurch Hospital, Romford, England
  - Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - North Staffs Royal Infirmary, Stoke-on-Trent, England
  - Royal Marsden Hospital, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - New Cross Hospital, Wolverhampton, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Velindre Hospital, Cardiff, Wales
  - Cumberland Infirmary, Carlisle
  - Saint Mary's Hospital, Portsmouth Hants
  - Royal Preston Hospital, Preston

REFERENCES:
- [Result] Hopwood P, Haviland JS, Sumo G, Mills J, Bliss JM, Yarnold JR; START Trial Management Group. Comparison of patient-reported breast, arm, and shoulder symptoms and body image after radiotherapy for early breast cancer: 5-year follow-up in the randomised Standardisation of Breast Radiotherapy (START) trials. Lancet Oncol. 2010 Mar;11(3):231-40. doi: 10.1016/S1470-2045(09)70382-1. Epub 2010 Feb 6. PMID 20138809
- [Result] Hopwood P, Haviland J, Mills J, Sumo G, M Bliss J; START Trial Management Group. The impact of age and clinical factors on quality of life in early breast cancer: an analysis of 2208 women recruited to the UK START Trial (Standardisation of Breast Radiotherapy Trial). Breast. 2007 Jun;16(3):241-51. doi: 10.1016/j.breast.2006.11.003. Epub 2007 Jan 19. PMID 17236771
- [Result] Venables K, Miles EA, Aird EG, Hoskin PJ; START Trial Management Group. The use of in vivo thermoluminescent dosimeters in the quality assurance programme for the START breast fractionation trial. Radiother Oncol. 2004 Jun;71(3):303-10. doi: 10.1016/j.radonc.2004.02.008. PMID 15172146